CLINICAL TRIAL: NCT05272423
Title: A Non-interventional, Non-treatment, Non-randomized, Single Coordinating Center, Decentralized Bio-specimen Collection Study in USA-based Adult Subjects With Acquired Resistance to KRAS Inhibitors
Brief Title: Studying Pathways of Resistance in KRAS-driven Cancers
Acronym: SPARK
Status: Active, not recruiting | Type: Observational
Sponsor: Addario Lung Cancer Medical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ALCMI-016
Record Dates: First submitted 2022-03-01; First posted 2022-03-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: KRAS P.G12C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood; archival tissue (optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1A: Patients who are currently progressing on a KRAS G12C inhibitor. Plasma for ctDNA analysis will be collected.
  Interventions: Diagnostic Test: FoundationOne® Liquid CDx
- Cohort 1B: Patients who have already had a sequencing assay performed to determine the resistance mechanism to a KRAS G12C inhibitor. These patients will be invited to share their data and medical history. Plasma for ctDNA analysis will be optional.
  Interventions: Diagnostic Test: FoundationOne® Liquid CDx

INTERVENTIONS:
Diagnostic Test: FoundationOne® Liquid CDx — The FoundationOne® Liquid CDx is an FDA-approved companion diagnostic that analyzes guideline-recommended genes from a simple blood draw.

SUMMARY:
Up to 250 patients from anywhere in the United States can remotely consent and participate to have plasma drawn locally and submitted to Foundation Medicine, Inc. (FMI), for the FoundationOne® Liquid Biopsy Assay. Patients who have had resistance mechanisms determined through other assays can also consent to share these data. The Investigator(s) will compare mechanisms of acquired resistance across drugs (e.g. sotorasib vs adagrasib) and between tumor types (e.g. NSCLC vs CRC) to determine if different resistance mutations arise in these settings.

DETAILED DESCRIPTION:
A hypothesis is that a remote participation plasma NGS study will characterize resistance mechanisms arising in KRAS-mutant cancers among individuals experiencing disease progression while on a KRAS-targeting therapy, and that subsequent therapies may be further personalized based on the results of plasma NGS testing.

After a web-based remote consent is obtained, subjects will be sent blood collection kits with the necessary materials for local draws and those specimens will be sent to the Dana-Farber Cancer Institute (DFCI), and rerouted to the central laboratory (Foundation Medicine, Inc.) for plasma NGS and to the ALCMI for storage. Plasma NGS results will be returned to the participant's treating physician, and the study team, aiming to be returned within approximately 2 weeks. In addition, subsequent treatments and clinical outcomes will be prospectively monitored. A correlation between the resistance mechanisms and clinical outcomes will be analyzed.

Patients with KRAS G12C mutant cancers will be enrolled in two cohorts.

* Cohort 1A will enroll patients who are currently progressing on a KRAS G12C inhibitor and plasma for ctDNA analysis will be collected from these patients remotely.
* Cohort 1B will enroll patients who have already had a sequencing assay performed to determine the resistance mechanism to a KRAS G12C inhibitor. These patients will be invited to share their data and medical history with the study team. Plasma for ctDNA analysis will be optional for this cohort.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1A- Liquid Biopsy

  1. Participants older than 18 years old at the time of consent or age of majority for residential state.
  2. Demonstration of having advanced KRAS G12C positive cancer.
  3. Systemic progression (not CNS only progression) within the past 30 days, having previously been treated with a therapeutic, targeting the specific KRAS mutation.
  4. Patient must not have started a new line of therapy before signing the informed consent form.
  5. Willingness to provide a blood specimen prior to the initiation of a new line of treatment.
  6. Willingness to provide clinical and medical information to the study team as required.
  7. Ability to read, write and communicate in English.
  8. Ability to sign a web-based informed consent form.

Cohort 1B- Data Sharing

1. Participants older than 18 years old at the time of consent or age of majority for residential state.
2. Demonstration of having advanced KRAS G12C positive cancer.
3. Systemic progression (not CNS only progression) after being treated with a therapeutic targeting the specific KRAS mutation.
4. Patient must have prior tumor genotyping available (tissue or plasma) after progression on therapeutic targeting the specific KRAS mutation.
5. Willingness to provide clinical and medical information to the study team as required.
6. Ability to read, write and communicate in English.
7. Ability of the participant or legally authorized representative (LAR) to sign a web-based informed consent form.

Exclusion Criteria:

1. Participants who are unable to comply with the study procedures.
2. Known existence of an uncontrolled intercurrent illness including, but not limited to, psychiatric illness or social situations that would impair compliance with study requirements.
3. Participants who have previously enrolled to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with a diagnosis of acquired resistance to KRAS inhibitors
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Genomic mechanisms of acquired resistance to KRAS inhibitors | up to 24 months follow-up
  The Investigator(s) will summarize mechanisms of acquired resistance with descriptive statistics (percentage and confidence interval), and compare across drugs (e.g., sotorasib vs adagrasib) and between tumor types (e.g., NSCLC vs CRC) to determine if different resistance mutations arise in these settings, using Fisher's exact test.

CONTACTS AND LOCATIONS:
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SPARK study webpage — https://alcmi.org/research/spark/